CLINICAL TRIAL: NCT06274372
Title: The Effect of Flow-controlled Ventilation on Hemodynamic and Respiratory Parameters in Laparoscopic Surgeries, Prospective Randomized Study
Brief Title: The Effect of Flow-controlled Ventilation on Hemodynamic and Respiratory Parameters in Laparoscopic Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nurseda Dundar, Principal Investigator, Derince Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FCV,V-2202
Record Dates: First submitted 2023-01-24; First posted 2024-02-23 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Laparoscopic Surgeries
Keywords: flow controlled ventilation; laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Other): patients ventilated with volume controlled ventilation
  Interventions: Device: volume controlled ventilation
- flow controlled ventilation (Experimental): patients ventilated with flow controlled ventilation
  Interventions: Device: flow controlled ventilation

INTERVENTIONS:
Device: flow controlled ventilation — effects of flow controlled ventilation
  Arms: flow controlled ventilation
Device: volume controlled ventilation — effects of volume controlled ventilation
  Arms: control group

SUMMARY:
It is aimed to investigate the effect of flow controlled ventilation on intraoperative respiratory parameters and hemodynamic parameters in laparoscopic operations.

DETAILED DESCRIPTION:
Study will begin after ethics committee approval and the patient's written and verbal consent .

Prospective observational studies will be conducted on patients over the age of 18 who will undergo laparoscopic surgery in the operating rooms. Patients who did not give verbal and written consent, emergency interventions, patients at risk of aspiration, patients with an ASA physical status above 3 and a diagnosis of COPD will be excluded.

Patients will be randomized and divided into two groups. Patients intraoperatively ventilated with a conventional ventilator (GE™ Avance™ CS2, VCV mode) Group 1, intraoperative ventilation Ventinova ( Evone®, Ventinova Medical, Eindhoven, the Netherlands, FCV mode) will be referred to as Group 2. Standard monitoring (ECG; SpO2, end tidal CO2,arterial blood pressure) will be applied to all patients. Anesthesia induction will be performed with propofol, fentanyl, rocuronium bromide as standard; In addition, anesthesia maintenance of the patients will be provided with propofol and remifentanil.

Respiratory parameters such as peripheral SpO2, PaCO2 value, peak airway pressure of each group will be recorded, and intraoperative hemodynamic parameters (systolic, diastolic, mean blood pressure, heart rate) of each group will be monitored and recorded.

Postoperative respiratory functions and length of hospital stay of all patients will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria: patients who will undergo laparoscopic surgeries, ASA 1,2,3 physical status

-

Exclusion Criteria:

* patients who do not give verbal and written consent, emergency interventions, patients at risk of aspiration, patients with an ASA physical status above 3 and a diagnosis of COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
effects of flow controlled ventilation on arterial pressure | intraoperatively
  Arterial blood pressure in mmHg
effectcs of flow controlled ventiletion on endtidal CO2 | intraoperatively
  endtidal CO2 in mmHg
effects of flow controlled ventilation on mean arterial pressure | intraoperatively
  mean arterial pressure change in percent
effects of flow controlled ventilation on heart rate | intraoperatively
  heart rate in bpm
effectcs of flow controlled ventiletion on peak airway pressure | intraoperatively
  peak airway pressure in cmH2O

SECONDARY OUTCOMES:
respiratory related complications | intraoperative period and postoperative first week
  rate of ventilator-associated pneumonia, rate of postoperative atelectasis, respiratory distress requiring reintubation by percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Nurseda Dundar, MD, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli Derince Training and Research Hospital, Derince, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No